CLINICAL TRIAL: NCT03360357
Title: Laparoscopic Vaginal Cuff Suturing Proficiency Following Two Standard Educational Approaches: A Randomized Controlled Trial
Brief Title: Laparoscopic Vaginal Cuff Suturing Profienciency for OBGYN Residents
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants to enroll.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher C. Destephano, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-008825
Record Dates: First submitted 2017-11-06; First posted 2017-12-04 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- guided drills (Experimental): These people will be going through all the guided drills before being evaluated.
  Interventions: Procedure: Guided drills
- Self-trained (No Intervention): These people will watch a video and be able to practice by themselves without having any direction regarding how and what to practice.

INTERVENTIONS:
Procedure: Guided drills — These residents will perform 5 set of exercises:
  1. "Needle Dance" (Learning to manipulate the suture)
  2. "Loopy Loop" (Learning to place needle through a loop)
  3. "Slalom Course" (Passing the needle and suture through 5 rings right handed and left handed)
  4. "Dense Matter" (Passing the needle through dense material without losing control of the needle)
  5. "Respect for tissue" (Passing the needle through flimsy material without tearing)
  Arms: guided drills

SUMMARY:
A recent survey of obstetrics and gynecology fellowship program directors showed that graduating OB/GYN residents may be underprepared for advanced laparoscopic training, necessitating an evaluation of the current structure of resident and fellow curriculum. Specifically, only 46% of first year fellows were able to independently perform an abdominal hysterectomy. Out of 28 residents tested using a previously validated laparoscopic cuff suturing model, only 8 (28.6%) passed the assessment.

For this reason, it is necessary to identify the most effective and efficient educational approaches to obtain procedural proficiency. Time and effort has been placed in developing simulation programs. Simulation has shown promising outcomes in improving the performance of trainees and attending physicians with the ultimate objective of generating better surgeons. A previous meta-analysis of simulation-based educational assessments demonstrated that these assessments correlate positively with patient-related outcomes. However, there are limited studies with adequate validity to use simulation for summative evaluations of performance for gynecology residents. The widely used Fundamentals of Laparoscopic Surgery (FLS) program is used for credentialing of general surgeons, however, a systematic review suggested that more validity evidence is required to support its content (selection of tasks and scoring rubric) and the consequences (favorable and unfavorable impact) assessment. Although there has been an increase in the number of models available to teach OB/GYN common gynecologic procedures, there is a lack of evidence to support that these methods are actually allowing residents to create better surgical skills.

To address the current limitations in OB/GYN training, the investigators have developed short, guided drills that cover the steps required for laparoscopic suturing and allow residents opportunities for deliberate practice. These drills will be tested compared to residents watching a laparoscopic suturing video and practicing using a high fidelity, suturing simulation model. Both of these methods are standard educational approaches for teaching laparoscopic skills, but it is unknown if one of the approaches is more effective than the other.

DETAILED DESCRIPTION:
Methods: Describe, in detail, the research activities that will be conducted under this protocol:

This study is a randomized controlled trial comparing laparoscopic suturing skills, specifically vaginal cuff closure, of OBGYN residents, fellows, and faculty using two different teaching methods and evaluate if there is any significant difference in their performance after teaching with the two different educational approaches. The laparoscopic camera/scope within a box trainer will video record the drills and the cuff suturing evaluation anonymously. These anonymous videos will be used to set proficiency standards for the drills and evaluate which educational approach is most effective.

The educational video and high fidelity simulation practice group will watch a 10 minute educational video on how to suture laparoscopically and then practice using a high fidelity simulation model for 15 minutes.

The second group is going to consist of "guided drills" as their laparoscopic training for 15 minutes. The residents will perform 5 set of exercises:

1. "Needle Dance" (Learning to manipulate the suture)
2. "Loopy Loop" (Learning to place needle through a loop)
3. "Slalom Course" (Passing the needle and suture through 5 rings right handed and left handed)
4. "Dense Matter" (Passing the needle through dense material without losing control of the needle)
5. "Respect for tissue" (Passing the needle through flimsy material without tearing)

After these exercises have been completed the participants will proceed to the 5 minute laparoscopic suturing evaluation. The evaluation will consist of closing the vaginal cuff in a previously validated simulator. The residents will have a determined amount of time to complete this task and the laparoscopic suturing will be filmed anonymously. Once the encounter is finished, the video will be saved, reviewed and graded using the previously validated global operative assessment of laparoscopic skills (GOALS).

* needle handling,
* getting the needle into the loop
* vaginal mucosa incorporation
* depth perception
* bimanual dexterity
* efficiency
* tissue handling
* Autonomy. Each area will consist of a score between 1 and 5. The "passing score" that defines proficiency will be 32 points as this number has been related to advance novice-expert in the past.

ELIGIBILITY:
Inclusion Criteria:

* Current OBGYN residents, fellows, and faculty at ACGME accredited residencies in the United States

Exclusion Criteria:

* - Non-current OBGYN residents at at ACGME accredited residencies in the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Proficiency of laparoscopic suturing of OBGYN residents | 15 minutes
  Vaginal cuff suturing proficiency will be higher in OB/GYN residents assigned to guided laparoscopic drills compared to residents assigned to an education video and high fidelity vaginal cuff suturing simulation model.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials